CLINICAL TRIAL: NCT03334500
Title: Evaluating in Vivo PARP-1 Expression With 18F-FluorThanatrace Positron Emission Tomography (PET/CT) in Prostate Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 13817
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ADP Ribose Transferases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Gleason 6 (n=10)
  Interventions: Device: [18F]FluorThanatrace; Drug: Poly(ADP Ribose) Polymerase 1
- Cohort 2 (Experimental): Gleason 7-8 (n=10)
  Interventions: Device: [18F]FluorThanatrace; Drug: Poly(ADP Ribose) Polymerase 1
- Cohort 3 (Experimental): Gleason 9 or oligometastic disease (n=10)
  Interventions: Device: [18F]FluorThanatrace; Drug: Poly(ADP Ribose) Polymerase 1

INTERVENTIONS:
Device: [18F]FluorThanatrace — Fluorine-18 labeled FluorThanatrace [18F]FTT can be synthesized with high specific activity so the quantity of mass injected with the radiopharmaceutical is < 10 μg.
  Other Names: 18F-FTT
Drug: Poly(ADP Ribose) Polymerase 1 — Poly(ADP-ribose) polymerase (PARP) is a family of enzymes involved in base excision repair (the repair of DNA single-strand breaks) and alternative end joining (repair of DNA double-strand breaks). The molecular basis of PARP1 inhibitor function may depend on the dual roles of PARP1 as a modulator of gene transcription in addition to DNA damage repair 3.
  Other Names: PARP 1

SUMMARY:
Men with a history of prostate cancer may be in this study. Subjects recommended for a prostatectomy or oligometastectomy will undergo PET/CT imaging using a novel radiotracer [18F]FTT to evaluate PARP-1 activity in known or suspected sites of primary or metastatic disease. Imaging will be compared with pathology results, including additional research assays when possible.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be ≥ 18 years of age
* Biopsy proven prostate cancer
* Must meet one of the following criteria:

  1. At least two tissue cores containing at least 50% tumor (per pathology report) OR
  2. At least one lesion that is 1 cm or greater in size by standard imaging (e.g. ultrasound, MRI, CT). Only one type of imaging is required to show a lesion of 1 cm or greater in order for the patient to be eligible to participate in this study.
* Recommended for clinically indicated radical prostatectomy or oligometastectomy
* Willing to allow use or collection of pathology tissue for the purposes of research from either clinical biopsy or surgical procedure (if adequate tissue is available)
* Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.

Exclusion Criteria:

* Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
* Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
* Only individuals (aged 18 or over) who can understand and give informed consent will be approached to participate in this study. Individuals who are considered to be mentally disabled will not be recruited for this study. All subjects must understand and be able to give informed consent. We will not be using specific methods to assess decisional capacity. Economically disadvantaged persons will not be vulnerable to undue influence, as this study offers no compensation. All individuals will be told that their choice regarding study participation will in no way change their access to clinical care. This should negate any undue influence or coercion. Women, children, fetuses, neonates, or prisoners are not included in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Dan Pryma, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No